CLINICAL TRIAL: NCT01630200
Title: Effects of ROFLUMILAST on Markers of Subclinical Atherosclerosis In Stable COPD; the ELASTIC-trial
Brief Title: Effects of ROFLUMILAST on Subclinical Atherosclerosis in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: ELASTIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LudwLudwig Boltzmann Institute for COPD and Respiratory Epidemiology (Network)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ELASTIC2011
Record Dates: First submitted 2012-06-04; First posted 2012-06-28 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-01

CONDITIONS: Chronic Obstructive Pulmonary Disease and Allied Conditions
Keywords: COPD; comorbidity; arterial stiffness; roflumilast
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Roflumilast (Active Comparator): Active arm including patients who receive the study drug (500µg Roflumilast once daily)
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator): Control arm including patients who receive the placebo tablet (once daily)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — Roflumilast coated tablet, 500µg oral application, once daily in the morning
  Other Names: Daxas
  Arms: Roflumilast
Drug: Placebo — Placebo coated tablet (visually identical to 500µg Roflumilast tablet), oral application, once daily in the morning
  Arms: Placebo

SUMMARY:
Chronic obstructive pulmonary disease is associated with a low grade systemic inflammatory process. Systemic inflammation is hypothesized to maintain cardiovascular morbidity and mortality in COPD. Early changes of vascular integrity can be detected via markers of subclinical atherosclerosis.

Selective Inhibition of phosphodiesterase subtype 4 describes a promising therapeutic option in COPD with beneficial impact on lung function and exacerbation rate. Moreover, an anti-inflammatory effect of phosphodiesterase-4 inhibition was confirmed by recent data.

The aim of this study is to assess the effects of the phosphodiesterase-4 inhibitor Roflumilast on firstly surrogates of subclinical atherosclerosis and secondly markers of systemic inflammation in the peripheral circulation of patients with stable chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Over 40 years of age
* Smoking history of at least 10 pack years
* Chronic obstructive pulmonary disease at Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage II - IV diagnosed according to standard criteria.
* History of at least one COPD exacerbation requiring systemic corticosteroid treatment or hospitalisation in the previous year

Exclusion Criteria:

* Insufficient compliance to study medication (≤70% of tablets used) during 4 weeks run-in period
* History of acute exacerbation 4 weeks prior to run-in period
* Diagnosis of alpha-1-antitrypsin deficiency
* Diagnosis of asthma
* Acute respiratory infections (e.g. pneumonia)
* Severe acute infectious diseases (e.g. active hepatitis, HIV)
* Lung cancer
* Bronchiectasis
* Interstitial lung disease
* Any other relevant lung disease
* Acute myocardial infarction
* Systolic left ventricular dysfunction
* Congestive heart failure New York Heart Association Functional Classification (NYHA) severity grade IV
* Haemodynamically significant cardiac arrhythmias or heart valve deformations
* Peripheral arterial occlusive disease
* Acute or chronic renal/hepatic failure
* Active malignancy
* Autoimmune disease
* Pregnant or breastfeeding women
* Women no using or not willing to use adequate contraceptive measures for the duration of the trial
* Hypersensitivity to study medication or placebo
* Severe psychiatric or neurological disorders or history of depression associated with suicidal ideation or behaviour
* Galactose intolerance, lactase insufficiency or glucose-galactose malabsorption

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Otto C Burghuber, M.D., Principal Investigator — Department for Respiratory and Critical Care Medicine, Otto Wagner Hospital, Vienna
Locations (1):
- Deparment for Respiratory and Critical Care Medicine, Otto Wangner Hospital, Vienna, Austria

REFERENCES:
- [Derived] Urban MH, Kreibich N, Gleiss A, Funk GC, Hartl S, Burghuber OC. Effects of roflumilast on arterial stiffness in COPD (ELASTIC): A randomized trial. Respirology. 2021 Feb;26(2):153-160. doi: 10.1111/resp.13914. Epub 2020 Jul 28. PMID 32725799

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Department of Respiratory and Critical Care Medicine in the Otto Wagner Hospital in Vienna and supporting centres (hospitals, outpatient clinics, respiratory specialists).
Pre-assignment Details: After inclusion, patients entered a 4 week, single-masked run-in period with placebo application. Given sufficient compliance to medication (≥70% of tablets) patients were randomized to receive either the study drug (Roflumilast 500 μg) or placebo in a double-masked manner.
Period: Overall Study
Arm/Group | Roflumilast | Placebo
Started | 40 | 40
Completed | 33 | 34
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.5 [61 to 69.5] | 64.5 [56 to 72] | 64.5 [57 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 16 | 38
  Male | 18 | 24 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 40 | 40 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Carotid Femoral-Pulse Wave Velocity at Month 6
Description: Carotid femoral-Pulse Wave Velocity (cf-PWV) will be measured non-invasively via applanation tonometry (AtCor Medical, Sydney, Australia). Wave propagation time will be calculated by the system software, using an ECG-gated reference frame. Aortic PWV is defined as the distance between two recording sites (i.e. common carotid- and femoral artery) divided by the wave propagation time.
Time Frame: baseline, month 6
Measure: Least Squares Mean (95% Confidence Interval); unit: meters per second (m/s)
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 33 | 34
meters per second (m/s) | 1.07 [0.98 to 1.17] | 0.99 [0.91 to 1.08]

2. Secondary Outcome: Change From Baseline in Reactive Hyperemia Index at Month 6
Description: Endothelial dysfunction will be assessed by Flow Mediated Dilation via the Endopat device. This validated system measures the pulse wave amplitudes at the tip of both index fingers. The dominant arm will be occluded for 5 minutes by a sphygmomanometric cuff. After cuff deflation the pulse wave amplitude will be assessed to finally calculate the ratio of pulse wave amplitude before and after cuff-induced hyperemia. The so called reactive hyperemia index represents endothelial dysfunction at the level of conduit as well as resistance vessels.
Time Frame: baseline, month 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Index
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 33 | 34
Index | 0.99 [0.88 to 1.11] | 1.02 [0.91 to 1.15]

3. Secondary Outcome: Change From Baseline in Augmentation Index at Month 6
Description: The curve of the peripheral pressure wave will be recorded from the radial artery. Augmentation index (Aix) will be calculated from the generated central aortic pressure waveform via pulse wave analysis function. To correct for respective influences, Aix will be adjusted for a heart rate of 75 bpm. Appropriate intra observer validity will be assured via an operator index ≥ 80.
Time Frame: baseline, month 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Index
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 33 | 34
Index | -1.11 [-5.33 to 3.11] | -1.99 [-6.12 to 2.14]

4. Secondary Outcome: Change From Baseline in Matrix Metalloproteinase-9
Description: Circulating levels of Matrix Metalloproteinase-9 (MMP-9) will be quantified from venous blood samples via Enzyme-linked Immunosorbent Assay
Time Frame: baseline, month 6
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 33 | 34
ng/ml | -143 [-370 to 84.6] | -77 [-301 to 147]

5. Secondary Outcome: Change From Baseline in Asymmetric Dimethylarginine at Month 6
Description: Circulating levels of Asymmetric dimethylarginine (ADMA) will be quantified from venous blood samples via Enzyme-linked Immunosorbent Assay
Time Frame: baseline, month 6
Measure: Least Squares Mean (95% Confidence Interval); unit: µmol/l
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 33 | 34
µmol/l | 0.97 [0.88 to 1.06] | 0.91 [0.83 to 1.00]

6. Secondary Outcome: Change From Baseline in Tumor Necrosis Factor-alpha at Month 6
Description: Circulating levels of Tumor Necrosis Factor-alpha (TNF-alpha) will be quantified from venous blood samples via Enzyme-linked Immunosorbent Assay
Time Frame: baseline, month 6
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 33 | 34
pg/ml | 0.95 [0.82 to 1.08] | 1.06 [0.92 to 1.22]

7. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second at Month 6
Description: Forced Expiratory Volume in 1 second (FEV1) will be measured via standardized Spirometry
Time Frame: baseline, month 6
Measure: Least Squares Mean (95% Confidence Interval); unit: % predicted
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 33 | 34
% predicted | 1.02 [0.96 to 1.08] | 1.01 [0.96 to 1.07]

8. Secondary Outcome: Change From Baseline in 6-Minute Walk Test at Month 6
Description: 6-Minute Walk Test (6MWT) will be assessed to quantify functional exercise capacity following the standardized protocol of the American Thoracic Society
Time Frame: baseline, month 6
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 33 | 34
meters | 59.2 [18.3 to 100] | 0.69 [-39.7 to 41.1]

9. Secondary Outcome: Change From Baseline in COPD Assessment Test at Month 6
Description: COPD Assessment Test (CAT) will be assessed to quantify patients disease related symptoms and to measure the impact of COPD on a patient's life, and how this changes over time. CAT is a standardised and validated patient questionaire comprising 8 distinct questions about different COPD-related symptoms. Each symptom is quantified by the patient on a numeric scale ranging from 0 to 5. Each symptom gives a number of points quantified as interval data without decimal places. The 8 different numbers of points are added to a total number expressed as the final points of the CAT score. The minimum achievable number of points is 0 and the maximum achievable number of points is 40. Higher values provide high symptoms and worse outcome, lower values provide low symptoms and better outcome.
Time Frame: baseline, month 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 33 | 34
units on a scale | 0.42 [-1.36 to 2.19] | 1.2 [-0.57 to 2.98]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Roflumilast | Placebo
All-Cause Mortality (participants affected / at risk) | 2/40 | 1/40
Serious Adverse Events (participants affected / at risk) | 13/40 | 9/40
Other Adverse Events (participants affected / at risk) | 27/40 | 22/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast (N=40) | Placebo (N=40)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bronchoscopic lung volume reduction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary nodule (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Diabetic vasculopathy (Vascular disorders) | 1 (1) | 0 (0)
Bronchoscopy for bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Death (unknown origin) (Investigations) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypercapnic decompensation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Polypectomy (Gastrointestinal disorders) | 0 (0) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast (N=40) | Placebo (N=40)
Weight loss (Gastrointestinal disorders) | 6 (6) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Common cold (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loss of appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cramps in upper/lower extremities (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1)
Influenca (Infections and infestations) | 0 (0) | 2 (2)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 14 (19) | 16 (24)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Herniated vertebral disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes